CLINICAL TRIAL: NCT00648453
Title: Effect of Plavix Treatment on NO Production Measured by Laser Doppler Method Referring to Endothelial Function in Patients With Severe Coronary Heart Disease
Brief Title: Effect of Plavix on NO (Nitrogen Monoxide) Production of the Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8564
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Peripheral Arterial Disease
Keywords: Fontain II-III stage
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel (Plavix)

SUMMARY:
To determine whether in the laser Doppler flowmetric parameters characteristic of endothelial dysfunction at patients with clinically manifest atherosclerosis any change can be detected at plavix (clopidogrel) treatment. Laser Doppler /LD/ measurement combined with iontophoresis evaluates the effect of acetylcholine /ACh/ /endothelium dependent/ and sodium nitroprusside /NSP/ /endothelium independent/ on the microcirculation of the skin

ELIGIBILITY:
Inclusion Criteria:

* Proven, peripheral arterial disease, Fontain II-III stage, patient submitted to secondary prophylactic thrombocyte aggregation inhibiting treatment
* Doppler index < 0,8

Exclusion Criteria:

* Hypersensitivity to the active ingredient or one of the components of the drug
* Active pathological bleeding, e.g. gastric ulcer, intracranial bleeding
* Pregnancy, breast-feeding
* Severe, known hepatic insufficiency
* Severe, known renal insufficiency

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2002-12; Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Change of the laser Doppler parameters measured after three months clopidogrel /75 mg/day/ treatment compared to the pre-treatment values. | 3 months

SECONDARY OUTCOMES:
Safety of clopidogrel /75 mg/day/ treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Eros, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Budapest, Hungary